CLINICAL TRIAL: NCT05444933
Title: OCTOPUS: An Observational, Non-interventional, Non-comparative, Retrospective, Multicentre Study in Patients With Advanced Renal Cell Carcinoma (aRCC) Who Initiated Cabozantinib in 2nd Line Under Real-life Setting in France.
Brief Title: A Study to Collect Pre-existing Data on the Administration of Cabozantinib in Participants With Advanced Renal Cell Carcinoma (aRCC) Who Initiated Cabozantinib in 2nd Line in a Real-life Clinical Setting in France.
Acronym: OCTOPUS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60000-454
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Sequencing post-cabozantinib: Participants treated by cabozantinib and who received another systemic therapy post-cabozantinib.
- Long responders: Participants treated by cabozantinib and who had a disease controlled (CR, PR or SDi during > 12 months after cabozantinib initiation with or without additional local treatment).
- Non-responders: Participants treated by cabozantinib and who had a progressive disease less than 3 months after cabozantinib treatment initiation.
- Cabozantinib & rechallenge: Participants treated by cabozantinib who received systemic therapy and/or had prolonged treatment-free interval (≥ 12 weeks) between two cabozantinib treatment periods. Participants with at least one cabozantinib rechallenge could be included in this subgroup.
- Cabozantinib & therapeutic schedules: Participants treated by cabozantinib and who needed 1/ a dose increase following disease progression and/or a prior reduction, Or 2/ had any dose reduction/dose interruption of cabozantinib (schedule adaptation).
- Cabozantinib & local treatment: Participants treated by cabozantinib and who needed concomitant local treatment (LT) by surgery or radiotherapy
- Cabozantinib & elderly patients: Participants treated by cabozantinib and aged ≥ 75 years

SUMMARY:
Cabozantinib is an orally bioavailable tyrosine kinase inhibitor (TKI) approved in patients with aRCC previously treated with a Vascular Endothelial Growth Factor (VEGF)-targeted therapy. Cabozantinib has been increasingly used in routine care in second line and more in advanced or metastatic RCC in France.

Cabozantinib effectiveness and safety notably in a real-word setting are now well known, but too many questions that arise during the routine care of patients with aRCC remain unanswered by the current literature.

Obtaining data on cabozantinib effectiveness and treatment pattern in those participants subpopulations will allow physicians to improve patients care.

The aims of this study are to describe the effectiveness - in terms of Duration of Treatment (DOT), Best Overall Response (BOR) and Progression-Free Survival (PFS) - and the safety of second line cabozantinib a real-life setting in France and to address the unanswered questions that arise during the routine care of patients with aRCC treated with cabozantinib in order to improve the care of these participants.

DETAILED DESCRIPTION:
Since 2018, cabozantinib has been increasingly used in routine care in second line and more in advanced or metastatic RCC in France.

Cabozantinib effectiveness and safety notably in a real-word setting are now well known, but too many questions that arise during the routine care of patients with aRCC remain unanswered by the current literature.

As an example, there is currently no real-world data on cabozantinib in elderly patients (≥ 75 years old); in patients with a systemic therapy after progression under cabozantinib (only one published monocentric retrospective study on 56 participants); or in long responder patients (with a disease controlled after > 12 months of cabozantinib). Obtaining data on cabozantinib effectiveness and treatment pattern in those patient subpopulations will allow physicians to improve patients care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 age at the time of cabozantinib initiation.
* Pathologically confirmed diagnosis of Renal Cell Carcinoma (RCC) considered as advanced at the time of cabozantinib initiation.
* Cabozantinib initiated from 1st March 2018 to 1st March 2021 for an advanced RCC.
* Cabozantinib initiated in 2nd line according to local Summary of Product Characteristics (SmPC).

Exclusion Criteria:

* Participant medical file without documented follow-up visits (post-cabozantinib initiation).
* Participant alive at study initiation who is opposed to data collection.
* Participant who died before study initiation and who was opposed to data collection for research purposes when alive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An estimated total of 300 participants with aRCC and who started cabozantinib in 2nd line between 1st March 2018 and 1st March 2021 is planned to be included. Participants will be enrolled from approximately 25 centers in France
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Duration of treatment (DOT) of cabozantinib | From baseline up to 18 months
  Defined as the time between first and last intake of cabozantinib treatment, regardless of the treatment discontinuation reason.

SECONDARY OUTCOMES:
Best Overall Response (BOR), until disease progression/recurrence | From baseline up to 18 months
  Defined as the proportion of participants achieving the best response among Complete Response (CR), Partial Response (PR), Stable Disease (SDi) or Disease Progression (DP), The method used for the assessment of response to treatment will be left at the discretion of the physician
Progression Free Survival (PFS). | From baseline up to 18 months
  Defined as the time from the date of first cabozantinib intake to the date of first documented progression reported by the investigator or death from any cause. Disease progression will be assessed by tumour response evaluation according to investigator assessment.
Incidence of all adverse events (AEs). | From baseline up to 30 days after cabozantinib last intake
  Whether they are serious/non-serious, related/unrelated experienced by the participants during cabozantinib treatment period(s).
Incidence of all Special Situations. | From baseline up to 30 days after cabozantinib last intake
  Whether they are serious/non-serious, related/unrelated experienced by the participants
Type of subsequent therapy | From baseline up to 18 months
  Will be described in terms of type, other TKI, Immuno-Oncology therapy (IO), mammalian Target Of Rapamycin (mTOR) inhibitors, other
DOT of subsequent therapy | From baseline up to 18 months
Starting dose of subsequent therapy | From baseline up to 18 months
Reasons for cabozantinib discontinuation | From baseline up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- France (27):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - Institut Sainte Catherine, Avignon
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - Centre Chirurgie Urinaire et d'Andrologie, Cabestany
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - APHP (Créteil), Créteil
  - Centre Hospitalier Annecy-Genevois, Épagny
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Polyclinique de Gentilly, Nancy
  - CHU Nice, Nice
  - APHP, Paris
  - APHP (Paris Grenelle), Paris
  - Institut Mutualiste Montsouris, Paris
  - Hospices civils de Lyon, Pierre-Bénite
  - CH Quimper, Quimper
  - CHU Reims, Reims
  - Hôpital Foch, Suresnes
  - Oncopole CHU Toulouse, Toulouse
  - CHRU Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers